CLINICAL TRIAL: NCT03572569
Title: Risk Stratification in Children and Adolescents With Primary Cardiomyopathy
Acronym: RIKADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Other Study IDs: A30127; 81Z3100331 (Other Grant/Funding Number: DZHK (German Centre for Cardiovascular Research))
Record Dates: First submitted 2018-06-01; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Primary Cardiomyopathy; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Left Ventricular Noncompaction; Restrictive Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: Pediatrics; Cardiomyopathy; Heart failure; Risk stratification; Family screening; Genetics
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Heart Failure

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA; tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index patients: Patients ≤18 years with primary cardiomyopathy
- First-degree family members: Parents and siblings of index patients

SUMMARY:
RIKADA is a prospective study performing systematic family screening including clinical and genetic testing in pediatric patients with primary cardiomyopathy and their first-degree relatives with the aim to facilitate risk stratification.

DETAILED DESCRIPTION:
RIKADA is a long-term prospective study performing in-depth phenotype and genotype characterization in children and adolescents with primary cardiomyopathy and their first-degree family members. Family screening contains complete cardiac work-up with medical history, physical examination, 12-lead-/Holter-electrocardiogram, cardiopulmonary exercise testing, echocardiography, cardiovascular magnetic resonance (CMR) and laboratory including genetic testing. The aim is to facilitate early identification of at-risk individuals and contribute to patient-specific follow-up and therapy regimes preventing progressive heart failure and arrhythmia in pediatric CMP.

ELIGIBILITY:
Inclusion Criteria:

1. Index patients:

   * Age ≤18 years
   * written informed consent of parents/legal guardians
   * diagnosis of primary cardiomypathy:
   * DCM: left ventricular (LV) systolic dysfunction and dilatation greater than two standard deviations (SD) above the mean of a normal population
   * HCM: LV hypertrophy and septal wall thickness above two SD
   * RCM: diastolic dysfunction and concordant atrial enlargement
   * LVNC: separation of the myocardium into a compacted (C) and a non- compacted (NC) layer with an NC/C ratio >2 in echocardiography and/or >2.3 in CMR
   * ARVC: according to the revised Task Force Criteria
2. First-degree family members (parents and siblings):

   * Age ≥3 years
   * written informed consent of parents/legal guardians and siblings ≥18 years

Exclusion Criteria:

* unwillingness to give consent
* myocardial inflammation / myocarditis
* systemic disease with cardiac involvement (secondary cardiomyopathy)
* structural congenital heart disease

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Department of pediatric cardiology including outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
major cardiovascular events | from date of enrollment until the date of death, mechanical circulatory support or heart transplantation, assessed up to 8 years
  death, need for mechanical circulatory support or heart transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Felix Berger, MD, Principal Investigator — German Heart Institute; Sabine Klaassen, MD, Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - German Heart Institute, Berlin

REFERENCES:
- [Derived] Al-Wakeel-Marquard N, Seidel F, Kuhnisch J, Kuehne T, Berger F, Messroghli DR, Klaassen S. Midwall Fibrosis and Cardiac Mechanics: Rigid Body Rotation Is a Novel Marker of Disease Severity in Pediatric Primary Dilated Cardiomyopathy. Front Cardiovasc Med. 2022 Feb 17;8:810005. doi: 10.3389/fcvm.2021.810005. eCollection 2021. PMID 35252369
- [Derived] Al-Wakeel-Marquard N, Degener F, Herbst C, Kuhnisch J, Dartsch J, Schmitt B, Kuehne T, Messroghli D, Berger F, Klaassen S. RIKADA Study Reveals Risk Factors in Pediatric Primary Cardiomyopathy. J Am Heart Assoc. 2019 Aug 6;8(15):e012531. doi: 10.1161/JAHA.119.012531. Epub 2019 Jul 23. PMID 31333075